CLINICAL TRIAL: NCT06376500
Title: Effects of Transcranial Direct Current Stimulation for Enhancing Cognitive Function in Individuals With Persistent Post-Concussion Syndrome: A Pilot fMRI/1H-MRS Study
Brief Title: Effects of tDCS for Enhancing Cognitive Function in Individuals With Persistent Post-Concussion Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Yvonne Han, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20240223001
Record Dates: First submitted 2024-04-08; First posted 2024-04-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-03

CONDITIONS: Transcranial Direct Current Stimulation; Post-Concussion Syndrome; Functional Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-tDCS (Experimental): For active-tDCS condition, participants will receive stimulation on the dorsolateral prefrontal cortex with ramp up and ramp down mode for 10 seconds, eliciting a tingling sensation on the scalp that fades over seconds.
  Interventions: Device: tDCS with cognitive training programme
- Sham-tDCS (Sham Comparator): For sham-tDCS condition, participants will receive initial stimulation with ramp up and ramp down mode for 30 seconds, eliciting a tingling sensation on the scalp then it will be discontinued.
  Interventions: Device: tDCS with cognitive training programme

INTERVENTIONS:
Device: tDCS with cognitive training programme — Participants will complete tDCS over 10 sessions in 2 weeks (once per day, for 10 consecutive working days), while performing the executive function training tasks. The training session will last for 20 minutes and it is comprised of 5 exercises targeting at information processing speed and executive function capacities. Each exercise lasts for approximately 4 minutes, totaling approximately 20 minutes.

SUMMARY:
Globally, 10 million new traumatic brain injury (TBI) cases are estimated annually, with mild traumatic brain injury (mTBI) accounting for 75-90% of all TBI cases. It is estimated that 40-80% of individuals with mTBI may experience the post-concussion syndrome (PCS), which is characterized by a range of physical, cognitive, and emotional symptoms. Although the underlying basis of cognitive dysfunction of patients with persistent PCS remains to be clarified, converging evidence shows that the clinical symptoms is underpinned by abnormal neural information processing as a result of axonal injury due to mTBI. Recent studies have demonstrated abnormalities in both structural and functional cortical connectivity, and a loss of cortical excitability-inhibitory (E/I) balance after TBI. Yet, there is no consensus for treating chronic symptoms of concussion, and PCS remains a chronic and highly disabling condition. One potential treatment option is transcranial direct current stimulation (tDCS), a non-invasive brain stimulation technique that has been shown to modify behavior by enhancing connectivity between targeted brain areas. However, research on the therapeutic effect of tDCS on PCS symptoms is limited, and the neurologic mechanisms underlying its effects are not well understood. The proposed study aims to address these knowledge gaps by examining the effects of tDCS on the central nervous system function in patients with PCS, with a specific focus on functional cortical connectivity and cognitive functions such as processing speed and executive function. The study also aims to add value to existing evidence by potentially opening new directions for designing intervention programs for the treatment of PCS after mTBI.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old or older;
* having a history of a mild TBI (less than 30 minutes loss of consciousness) 1-6 years prior to the study;
* able to communicate in Chinese.

Exclusion Criteria:

* being without a confirmed diagnosis from the medical practitioner;
* having a history of other neurological and psychiatric disorders, skull defect, recent medical instability (within 3 weeks);
* being pregnant;
* being medication for a psychiatric condition (e.g., major depression, anxiety, schizophrenia);
* with any implanted devices or suffering from real claustrophobia or feel uncomfortable in small, enclosed spaces, like MRI tunnel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Average standardised score of executive function tests | First day of intervention, 1 day after the last day of intervention (2 time points, up to 2 weeks)
  The executive function of the PCS subjects will be assessed using the Executive Composite score, which combines scores from various executive function tests.Simple-task processing speed will be evaluated using the CANTAB® 5-choice Reaction Time (RTI) task, which measures the ability to focus on relevant information while ignoring distractions. It requires participants to react as soon as a yellow dot appears on screen. Complex-task processing speed will be assessed using the computerized version of the Wisconsin Card Sorting Test (WCST), which assesses cognitive flexibility. The test requires subjects to correctly match the response cards with several stimulus cards according to feedback provided based on a rule. The mean reaction time is calculated for the trials giving a correct answer during WCST. The reaction time measured from both tasks will be converted to standard scores and averaged to yield an executive composite score. Lower scores indicate poorer executive functioning.

SECONDARY OUTCOMES:
Change in CANTAB® cognitive test - Reaction Time (RTI) | First day of intervention,1 day after the last day of intervention (2 time points, up to 2 weeks)
  RTI assesses motor and mental response speeds, reaction time, response accuracy and impulsivity. It consists of 30 trials with five potential targets and requires participants to make flexible responses as fast as possible to the target stimulus (shown in yellow). Specifically, movement and reaction time will be measured, where shorter duration reflects faster processing speed.
Change in CANTAB® cognitive test - Multitasking Test (MTT) | First day of intervention,1 day after the last day of intervention (2 time points, up to 2 weeks)
  MTT assesses the ability to resolve the interference of task-irrelevant information (stroop-like effect). The test displays an arrow which can appear on either the left or right side of the screen and can point to either the left or right side. In each trial, participants are presented with a cue that indicates which button to press according to two different rules. And the rules that participants have to follow may change from trial to trial in a randomized order. Participant's response latencies and error scores will be measured.
Change in CANTAB® cognitive test - Spatial Working Memory (SWM) | First day of intervention,1 day after the last day of intervention (2 time points, up to 2 weeks)
  SWM assess the memory ability of visuospatial information. Participants are required to search the tokens from a number of boxes but not pressing the boxes which tokens have been found. Errors (lower scores indicate lower repetition on pressing the same boxes that token has been found) and strategy (lower scores suggest higher strategy use in begin of choosing the same boxes) will be measured.

OTHER OUTCOMES:
Exploratory mediator - default mode network (DMN) activation | First day of intervention,1 day after the last day of intervention (2 time points, up to 2 weeks)
  The DMN activation, indexed by fMRI resting state data will be assessed. Neuroimaging data will be acquired from the whole brain using a 64-channel head coil on a 3T Siemens MRI scanner. Resting-state data will be registered to each participant's high-resolution structural image and then normalized into the standard Montreal Neurological Institute (MNI) space. Mediation analyses will be performed to determine if the enhanced network organization in PCS patients, as indexed by DMN activation, will mediate the beneficial effect of tDCS
Exploratory mediator - excitability-inhibitory (E/I) ratio | First day of intervention,1 day after the last day of intervention (2 time points, up to 2 weeks)
  The E/I ratio, indexed by MRS data will be assessed. The MRS acquisition protocol is adopted from Sapey-Triomphe and the colleagues. Magnetic resonance spectra will be acquired using the Hadamard Encoding and Reconstruction of MEGA-Edited Spectroscopy (HERMES) sequence, allowing for simultaneous quantification of GABA + and Glx (glutamine and glutamate). The MRS acquisition parameters will be set as follows: 320 averages, TR = 2000 ms, TE = 80 ms, 2048 data points, 2000 Hz spectral width, MOIST water suppression, 90°excitation/180°refocusing pulses, 20 ms editing pulses at frequencies 1.9 ppm for GABA. Interleaved Water Reference correction will be used to limit the effect of scanner drift. Twenty unsuppressed water reference scans (at TE = 80 ms) will also be acquired. Mediation analyses will be performed to determine if the enhanced network organization in PCS patients, as indexed by E/I balance, will mediate the beneficial effect of tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Han, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hung Hom, Kowloon, Hong Kong